CLINICAL TRIAL: NCT01422447
Title: Prevention and Mental Health Education for Mental Health Problems in Community: A Model of Common Mental Health Problems in Seven Metropolis of China
Brief Title: Research of Prevention and Intervention of Mental Health Problems
Acronym: RPIMHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MZhao-001
Record Dates: First submitted 2011-08-18; First posted 2011-08-24 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Anxiety; Depression; Alcohol-abuse
Keywords: mental health education; community-based
MeSH Terms: conditions — Anxiety Disorders; Depression; Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- community intervention (Experimental): Feedback on assessment results: distribute relevant brochures and hold regular lectures on depression, anxiety and alcohol-abuse.
  Interventions: Other: community intervention
- regular intervention control (Active Comparator): the subjects in the control group live in the used model
  Interventions: Other: regular intervention

INTERVENTIONS:
Other: regular intervention — the subjects in the control group live in the used model
  Arms: regular intervention control
Other: community intervention — in addition to regular intervention, those subjects in the intervention group will be given education intervention.
  Arms: community intervention

SUMMARY:
The purpose of this research is to establish a suitable community-based model for Chinese culture,to improve the community recognition of common mental disorders,as well as its treatment and control.

DETAILED DESCRIPTION:
The project will select seven metropolis,through multi-center collaborative research,use of interdisciplinary methods and combining qualitative and quantitative research methods.Community resources will be integrated so as to build the Chinese model of community mental health services and to establish the routine for common mental disorders. Evaluation criteria for community mental health needs to be developed for the process of health education and intervention techniques.

ELIGIBILITY:
Inclusion Criteria:

1. general population: 13-65-year-old,
2. high-risk groups: not yet shown symptoms of mental disorders, but exposed to epidemiological risk factors for anxiety,depression and alcohol abuse.A part may be at risk for future depression,anxiety and alcohol abuse,for example: post-disaster population,Stress-related groups, the unemployed and laid-off people, high risk of psychological disorders (chronic treatment of various medical institutions and disabled, the mentally ill family members).
3. early stage of mental disorders in population:the subjects have the problem of depression, anxiety or alcohol abuse, but not yet diagnosed with depression, anxiety disorders or alcohol abuse.

Exclusion Criteria:

those who have been diagnosed with depression,anxiety or alcohol abuse and other psychiatric disorders will be excluded from this study.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42016 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
evaluate the changes of mental health state of community residents before and after intervention | 12 months
  we will use several scales such as SRHMS,SE,SEI,PSS,SCSQ,PHQ,AUDIT,scale of mental health knowledge and attitude survey and suicide related problems to evaluate the effect of our intervention.

SECONDARY OUTCOMES:
prevalence of depression,anxiety and alcohol abuse | 12 months
  use scales of PHQ-9,PHQ-7 and AUDIT to investigate prevalence of depression,anxiety and alcohol abuse.
public awareness and attitude towards mental health knowledge | 12 months
  designed related questionnaires to investigate the public's awareness and attitude towards mental health knowledge.
service needs and utilization | 12 months
  use qualitative research methods to ivestigate service needs and utilization of three target population in community.
the reliability and validity of PHQ-9, HPQ-7 and AUDIT | 6 months
  use MINI as the gold standard to evaluate the reliability and validity of PHQ-9, HPQ-7 and AUDIT in community and university students
assessment of the situation of community mental health service resources | 1 month
  we use scales to evaluate the situation of community mental health service resources
assessment the changes of early stage of mental disorders in population before and after intervention | 3 months
  we will use several sacles such as assessment scale of motivation changes,alclhol behavior and willingness and confidence of abstain from drinking to evaluate the changes before and after intervention with people who have alcohol abuse problems and use SAS,SDS and IBS to evaluate the changes in people who have depression and anxiety problems.

CONTACTS AND LOCATIONS:
Overall Officials: Min ZHAO,, Ph.D., Principal Investigator — Shanghai Mental Health Center
Locations (7):
- China (7):
  - Capital Normal University, Beijing, Beijing Municipality
  - Shenzhen mental health center, Shenzhen, Guangdong
  - Mental Health Center in Hunan Province, Hunan, Hunan
  - Harbin medical university, Harbin, Jilin
  - 中国, Shanghai, Shanghai Municipality
  - Mental Health of Sichuan Province, Sichuan, Sichuan
  - Mental Health of Xinjiang Province, Xinjiang, Xinjiang